CLINICAL TRIAL: NCT02413554
Title: Rivastigmine Patch Effect on the Post-operative Delirium Limited to Femur Neck Fracture Operation in Patients at Risk of Dementia.
Brief Title: Rivastigmine Patch Effect on the Post-operative Delirium in Patients at Risk of Dementia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Youn Young Chul, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NR0001
Record Dates: First submitted 2015-04-02; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Delirium
Keywords: acetylcholinesterase inhibitors; rivastigmine patch; post-operational delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patch applied patients (Experimental): The investigators had enrolled consecutively the patients who were going to operation after femur neck fracture.
  Participants were applied the 5 unit rivastigmine patches from 3 days before and 7 days after the femur neck operation.
  Interventions: Drug: Rivastigmine patch
- Patch non-applied patients (No Intervention): The participants who were going to operation after femur neck fracture were not applied the rivastigmine patches.

INTERVENTIONS:
Drug: Rivastigmine patch — acetylcholine esterase inhibitor
  Other Names: exelon patch
  Arms: Patch applied patients

SUMMARY:
Delirium is a common and serious condition and is associated with adverse outcome. The elderly who have cognitive dysfunction are expected to show delirium more frequently. It is most likely that delirium represents a response to impaired cholinergic neurotransmission. Investigators aimed to establish the preventive effect of the cholinesterase inhibitor, rivastigmine patch, on the post-operative delirium limited to femur neck fracture operation in patients at risk of dementia.

DETAILED DESCRIPTION:
Investigators evaluated the delirium prevention effect of rivastigmine patch in patients with femur neck fracture and cognitive impairment. Investigators measured the frequency and severity of post-operation delirium in the patch applied and non-applied subjects.

ELIGIBILITY:
Inclusion Criteria:

* Consecutively enrolled the patients who is going to operation after femur neck fracture.
* Patients agree to the informed consent.

Exclusion Criteria:

* depressive mood and their geriatric depression scale is over 6 / 15.
* Their Korean version MMSE(minimental status examination) are over 25, or global dementia scale (GDS) are under 3 or over 5.
* any delirious state at pre-operation period by DSM IV and CAM (Confusion Assessment Method)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the number of participants with delirium | up to 7th days
  investigators evaluated the delirium frequency in rivastigmine applied participants comparing with non-applied participants.

SECONDARY OUTCOMES:
delirium severity using delirium rating scale | up to 7th days
  to compare the severity of delirium in rivastigmine patch applied participants with non-applied

CONTACTS AND LOCATIONS:
Overall Officials: Young Chul Youn, MD, PhD, Principal Investigator — Dept of Neurology, Chung-Ang University Hospital